CLINICAL TRIAL: NCT03180528
Title: A Phase 2 Open-Label, Single-Arm Trial of the Efficacy of Topical Remetinostat on Basal Cell Carcinoma in Patients
Brief Title: Topical Remetinostat in Treating Patient With Cutaneous Basal Cell Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kavita Sarin (Other)
Collaborators: Medivir (Industry); National Institutes of Health (NIH) (NIH); American Skin Association (Other)
Responsible Party: Sponsor-Investigator, Kavita Sarin, Principal Investigator, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-40947; NCI-2017-00981 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); SKIN0037 (Other: Stanford)
Record Dates: First submitted 2017-06-06; First posted 2017-06-08 (Actual); Results first posted 2021-01-05 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-05

CONDITIONS: Skin Basal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Basal Cell | interventions — remetinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (remetinostat) (Experimental): Patients receive topical remetinostat 1% gel applied TID directly to the lesion, for 6 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Remetinostat

INTERVENTIONS:
Drug: Remetinostat — Applied topically under bandage occlusion
  Other Names: suberohydroxamic acid phenyl ester (SHAPE); SHAPE Gel; SHP 141; and 4 [[8 (hydroxyamino) 1,8 dioxooctyl]oxy] benzoic acid methyl ester

SUMMARY:
This phase 2 trial studies how well remetinostat works in treating patients with skin basal cell cancer. Remetinostat may slow the growth of basal cell cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Overall response rate of basal cell carcinoma (BCC) in subjects at 6 weeks.

SECONDARY OBJECTIVES:

I. Suppression of GLI1 (glioma-associated oncogene) expression in treated BCCs as compared with baseline.

II. Safety assessment of Remetinostat after 6 weeks of topical treatment.

OUTLINE:

Tumors receive Remetinostat topically three times per day (TID) for 6 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed for at least 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Must have at least one BCC lesion > 1 cm (BCC > 5 mm) in non-cosmetically sensitive site(s)
* Must be willing to apply the topical remetinostat 3 times daily for 6 weeks
* For women of child bearing potential, a negative urine pregnancy test
* Women of child bearing potential are expected to use an effective method of birth control while participating in the study and for 1 month after applying the last dose
* For male subjects with female partners of childbearing potential, agreement to use adequate contraception while participating in the study and for 1 month after applying the last dose
* Has signed and dated the current Institutional Review Board (IRB) approved informed consent document

Exclusion Criteria:

* Taking any medication known to interact with histone deacetylase (HDAC) inhibitors, such as valproate or anticoagulants
* Taking any medication known to affect hedgehog (HH) signaling pathway such as itraconazole
* Within the past 6 months, has used topical or systemic therapies that might interfere with the evaluation of the study medication during the study; specifically, these include the topical use to the study tumors of:

  * Glucocorticoids
  * Retinoids either systemically or topically (eg, etretinate, isotretinoin, tazarotene, tretinoin, adapalene)
  * Alpha hydroxy acids (eg, glycolic acid, lactic acid) to > 5% of the skin
  * 5 fluorouracil or imiquimod and/or
  * Itraconazole
* Has received treatment with systemic chemotherapy or agents known to be inhibitors of HH signaling, within 60 days to starting study medication
* Currently receiving systemic medications that could affect BCC tumors (eg, oral retinoids) or might interact with remetinostat
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, recurrent seizure history or psychiatric illness/social situations that would limit compliance with study requirements
* Moderate to severe immunosuppression due to disease or medication
* Known or previous hypersensitivity to histone deacetylase inhibitor (HDACi)
* History of congestive heart failure; cardiac arrhythmias; or other findings of ventricular dysfunction
* History of current evidence of malabsorption or liver disease
* Pregnancy or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-07-07 (Actual); Primary Completion 2020-07-07 (Actual); Study Completion 2020-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kavita Sarin, Principal Investigator — Stanford University
Locations (1):
- Stanford University, School of Medicine, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Remetinostat)
Started | 30
Completed | 27
Not Completed | 3
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1
Not completed — Eligible and enrolled, but withdrawn due to abnormal baseline laboratory values. | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Remetinostat)
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 21
  >=65 years | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.26 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 27
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 27
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Overall response is defined as achieving either a complete response (CR) or a partial response (PR). Response is based on the Response Evaluation Criteria in Solid Tumors (RECIST), as follows.
  * CR = tumor lesion becomes undetectable
  * PR = ≥30% decrease in total tumor diameter
  * Overall response (OR) = CR+PR
  * Stable Disease (SD) = decrease in total tumor diameter is >0% and <30%
  * Progressive Disease (PD) = increase in total tumor diameter Exact binomial 90% confidence intervals (90%) will be computed for OR. The data are reported accord to the per protocol analysis, ie, including lesions for subjects who were <70% compliant with drug treatment. For subjects who were compliant but dropped out, data from their last study visit will be used if they contribute a biopsy. The analysis population will include the participants who have provided pre-treatment and post-treatment biopsies. The outcome is reported as the percent of tumor lesions that achieve OR, with 90% CI.
Time Frame: At 6 weeks
Population: Analysis is on a per-lesion basis, and not a per-participant basis. Per protocol, analysis does not include lesions from participants <70% compliant with treatment regimen.
Measure: Number (90% Confidence Interval); unit: percentage of tumor lesions
Units Other Than Participants: Tumor lesions
Arm/Group | Treatment (Remetinostat)
Number analyzed (Participants) | 25
Number analyzed (Tumor lesions) | 33
percentage of tumor lesions | 69.7 [54.0 to 82.5]

2. Secondary Outcome: Number of Participants With a Decrease in Expression of the Hedgehog Biomarker Gene GLI1
Description: The effect of topical remetinostat gel 1% on decreasing expression of Hedgehog biomarker gene GLI1 was determined using the RNeasy Fibrous Tissue Mini Kit (Qiagen, Valencia, CA), a polymerase chain reaction (PCR) test kit. The levels observed at baseline and after 6 weeks treatment were obtained. The outcome is reported as the number of subjects for whom a decrease in expression of the Hedgehog biomarker gene GLI1 was observed, a number without dispersion.
Time Frame: 6 weeks
Population: Results are reported for those participants for whom baseline and 6-week analysis data were available. The COVID-19 epidemic adversely affected the ability of the laboratory to process and return results.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Remetinostat)
Number analyzed (Participants) | 6
Participants | 5

3. Secondary Outcome: Adverse Events Contributing to Treatment Discontinuation or Interruption
Description: Adverse events (AEs) contributing to treatment discontinuation or interruption are reported as the number of such events, a number without dispersion.
Time Frame: 6 weeks
Population: The outcome is reported as a number of adverse events (AEs), not as a number of participants. For some participants, multiple AEs contributing to treatment decisions.
Measure: Number; unit: adverse events
Arm/Group | Treatment (Remetinostat)
Number analyzed (Participants) | 29
adverse events
  AEs contributing to treatment interruption | 9
  AEs contributing to treatment discontinuation | 3

4. Secondary Outcome: Participants Who Discontinued Treatment or Had Treatment Interruption
Description: The number of participants who discontinued treatment or experienced treatment interruption within the first 6 weeks of treatment are reported as the number of such participants, a number without dispersion.
Time Frame: 6 weeks
Population: For some participants, multiple AEs contributing to the treatment decision.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Remetinostat)
Number analyzed (Participants) | 29
Participants
  Participants who experienced treatment interruption | 5
  Participants who discontinued treatment | 3

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Data are reported for subjects that received the study treatment only. Subjects who were enrolled, but were withdrawn without receiving study treatment due to abnormal baseline laboratory values are not included.
Arm/Group | Treatment (Remetinostat)
All-Cause Mortality (participants affected / at risk) | 0/29
Serious Adverse Events (participants affected / at risk) | 0/29
Other Adverse Events (participants affected / at risk) | 29/29
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Remetinostat) (N=29)
Eczema (Skin and subcutaneous tissue disorders) | 27 (27)
Pain of Skin (Skin and subcutaneous tissue disorders) | 6 (6)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (1)
Skin Ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, tumor hemorrhage (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-10-02): https://cdn.clinicaltrials.gov/large-docs/28/NCT03180528/Prot_SAP_001.pdf
  • Informed Consent Form (2020-04-15): https://cdn.clinicaltrials.gov/large-docs/28/NCT03180528/ICF_000.pdf